CLINICAL TRIAL: NCT00638235
Title: A Prospective, Multi-Center Study to Assess the AMS Pelvic Floor Repair System Devices for Prolapse Repair
Brief Title: Pelvic Floor Repair Systems for Prolapse Repair
Acronym: PROPEL
Status: Completed | Type: Observational
Sponsor: ASTORA Women's Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 1004; NCT00793039 (obsolete NCT alias)
Record Dates: First submitted 2008-02-28; First posted 2008-03-19 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic floor repair; prolapse; mesh
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- Phase I (IntePro, US only): AMS Apogee™ with IntePro(Began May 2006 - Closed)
  Interventions: Device: AMS Apogee™ with IntePro
- Phase I (InteXen LP, US only): AMS Apogee™ with InteXen LP (Began May 2006 - Closed)
  Interventions: Device: AMS Apogee™ with Intexen LP
- Phase II (France only): AMS Perigee™ with IntePro (Began February 2007 - Closed)
  Interventions: Device: AMS Perigee™ with IntePro
- Phase III/IV (Perigee IntePro Lite, US only): AMS Perigee™ with IntePro Lite (Began April 2007 - Closed)
  Interventions: Device: AMS Perigee™ with IntePro Lite
- Phase III/IV (Apogee IntePro Lite, US only): AMS Apogee™ with IntePro Lite (Began April 2007 - Closed)
  Interventions: Device: AMS Apogee™ with IntePro Lite
- Phase V (Elevate Posterior IntePro Lite, US & EU): AMS Elevate™ Apical & Posteiror with IntePro Lite (Began April 2008 - Closed)
  Interventions: Device: AMS Elevate™ Apical & Posteiror with IntePro Lite
- Phase V (Elevate Posterior InteXen, US only): AMS Elevate™ Apical & Posteiror with IntXen LP (Began April 2008 - Closed)
  Interventions: Device: AMS Elevate™ Apical & Posteiror with IntXen LP
- Phase VI (Elevate Anterior Gen 1, For Study Use Only, EU only): AMS Elevate™ Anterior & Apical with IntePro Lite (Generation 1, For Study Use Only, Began October 2008 - Closed)
  Interventions: Device: AMS Elevate™ Anterior & Apical with IntePro Lite (Gen 1, For Study Use Only)
- Phase VII (Elevate Anterior Gen 2, US & EU): AMS Elevate™ Anterior & Apical with IntePro Lite (Generation 2, Began April 2009 - Closed)
  Interventions: Device: AMS Elevate™ Anterior & Apical with IntePro Lite (Gen 2)

INTERVENTIONS:
Device: AMS Apogee™ with IntePro — Mesh implant for posterior wall pelvic organ prolapse
  Groups: Phase I (IntePro, US only)
Device: AMS Apogee™ with Intexen LP — Graft implant for posterior wall pelvic organ prolapse
  Groups: Phase I (InteXen LP, US only)
Device: AMS Perigee™ with IntePro — Mesh implant for anterior wall pelvic organ prolapse
  Groups: Phase II (France only)
Device: AMS Perigee™ with IntePro Lite — Mesh implant for anterior wall pelvic organ prolapse
  Groups: Phase III/IV (Perigee IntePro Lite, US only)
Device: AMS Apogee™ with IntePro Lite — Mesh implant for posterior wall pelvic organ prolapse
  Groups: Phase III/IV (Apogee IntePro Lite, US only)
Device: AMS Elevate™ Apical & Posteiror with IntePro Lite — Mesh implant for apical and posterior wall pelvic organ prolapse
  Groups: Phase V (Elevate Posterior IntePro Lite, US & EU)
Device: AMS Elevate™ Apical & Posteiror with IntXen LP — Graft implant for apical and posterior wall pelvic organ prolapse
  Groups: Phase V (Elevate Posterior InteXen, US only)
Device: AMS Elevate™ Anterior & Apical with IntePro Lite (Gen 1, For Study Use Only) — Mesh implant for anteiror and apical wall pelvic organ prolapse
  Groups: Phase VI (Elevate Anterior Gen 1, For Study Use Only, EU only)
Device: AMS Elevate™ Anterior & Apical with IntePro Lite (Gen 2) — Mesh implant for anteiror and apical wall pelvic organ prolapse
  Groups: Phase VII (Elevate Anterior Gen 2, US & EU)

SUMMARY:
1. This is a prospective, multi-center, post market study, which will be conducted under a common protocol.
2. The primary objective of the study is to evaluate long-term efficacy of the AMS Pelvic Floor Repair System devices for prolapse repair.
3. The study population is female subjects > 21 years of age who require surgical reconstruction of their pelvic floor due to prolapse.
4. The clinical data will be analyzed by comparing post-treatment data with the baseline data, with the subject acting as her own control. The follow-up is for two years after the procedure.
5. Prolapse improvement measured by ICS POP-Q Stage at 12-months will be the primary endpoint of the study. The secondary endpoints include quality of life changes from baseline and adverse event rates.

ELIGIBILITY:
Inclusion Criteria:

-Have been diagnosed with one or more clinically significant anterior, apical or posterior genital prolapse disorder(s) (symptomatic POP-Q stage II or higher) requiring surgical repair

Exclusion Criteria:

* The Investigator determines the subject is not a candidate for surgical repair of her genital prolapse.
* Subject has had a prior prolapse implant/procedure (i.e., IVS tunneler, Perigee, Apogee, graft augmented repair, etc) Note: previous traditional repairs are allowed.
* Subject has active or latent systemic infection or signs of tissue necrosis.
* Subject has restricted leg motion (inability to abduct or adduct leg positioning in the lithotomy position) with or without a hip replacement/prosthesis.
* Subject is currently pregnant or intends to become pregnant during the study period. Note: the risks and benefits of performing the procedure if the subject is planning future pregnancies should be carefully considered.
* Subject has had radiation therapy to the pelvic area.
* Subject has pelvic cancer, has had pelvic cancer within the past 12 months or has been on cytostatic medication within the past 12 months.
* Subject has a known hypersensitivity to the graft material(s).
* Subject has uncontrolled diabetes.
* Subject is on any medication which could result in compromised immune response, such as immune modulators.
* Subject was involved in any other research trial < 30 days of enrollment into this study.
* Subject has undergone previous pelvic surgery < 6 months prior to enrollment in this study.
* Subject is unwilling or unable to give valid informed consent.
* Subject is unwilling or unable to comply with the requirements of the protocol, complete all Quality of Life questionnaires and return for all follow-up visits.
* Subject is contraindicated based on intended use and warnings in the AMS PFR System devices for prolapse repair Instructions for Use (IFU).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult females ages > 21 years old requiring surgical repair of their genital prolapse
Sampling Method: Non-Probability Sample
Enrollment: 725 (Actual)
Dates: Start 2006-05; Primary Completion 2011-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Lukban, DO, Principal Investigator — Eastern Virginia Medical School
Locations (28):
- United States (17):
  - Kaiser Permanente - Dept. of Obstetrics & Gynecology, Downey, California
  - Institute for Women's Health & Body, Wellington, Florida
  - Atlanta Medical Research Institute, Alpharetta, Georgia
  - Rosemark Womencare Specialists, Idaho Falls, Idaho
  - Fore River Urology, Portland, Maine
  - Maine Medical Partners, Portland, Maine
  - Female Pelvic Health, Whitinsville, Massachusetts
  - Female Pelvic Medicine and Urogynecology Inst. of Michigan, Grand Rapids, Michigan
  - Michigan Medical P.C., Grand Rapids, Michigan
  - Women's Health Care Specialists, PC, Paw Paw, Michigan
  - Metro Urology, Plymouth, Minnesota
  - Piedmont Urology Associates, Gastonia, North Carolina
  - Huey & Weprin Obstetrics & Gynecology, Englewood, Ohio
  - South Carolina OB/GYN, Columbia, South Carolina
  - University of Tennessee - Dept of Obstetrics & Gynecology, Memphis, Tennessee
  - Texas Tech University Health Science Center - OB/GYN Department, El Paso, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
- UZ Leuven Dept of Urology, Leuven, Belgium
- France (5):
  - CMC Beau Soleil, Montpellier
  - Service urologie de Paris l'Hôpital Tenon, Paris
  - Hopital Cochin - Saint-Vincent de Paul - Groupement hospitalier universitaire Ouest, Paris
  - CHU de Rouen - Pavillon Derocque - Rez de Chaussée, Rouen
  - Clinique Adassa, Strasbourg
- Germany (2):
  - Dr. Rainer Lange, Alzey
  - Beckenbodenzentrum Munich, Munich
- University of Amsterdam, Academic Medical Center - Department of Gynaecology and Obstetrics, Amsterdam, Netherlands
- Hospitalet General de l'Hospitalet, Barcelona, Spain
- University Hospital of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lukban JC, Roovers JP, Vandrie DM, Erickson T, Zylstra S, Patel MP, Moore RD. Single-incision apical and posterior mesh repair: 1-year prospective outcomes. Int Urogynecol J. 2012 Oct;23(10):1413-9. doi: 10.1007/s00192-012-1692-4. Epub 2012 Mar 15. PMID 22419354
- [Result] Lukban JC, Beyer RD, Moore RD. Incidence of extrusion following type I polypropylene mesh "kit" repairs in the correction of pelvic organ prolapse. Obstet Gynecol Int. 2012;2012:354897. doi: 10.1155/2012/354897. Epub 2011 Dec 10. PMID 22190952
- [Result] Moore RD, Lukban JC. Comparison of vaginal mesh extrusion rates between a lightweight type I polypropylene mesh versus heavier mesh in the treatment of pelvic organ prolapse. Int Urogynecol J. 2012 Oct;23(10):1379-86. doi: 10.1007/s00192-012-1744-9. Epub 2012 May 10. PMID 22572917
- [Derived] Liedl B, Barba M, Wenk M. [Pelvic floor reconstruction-update 2024: prolapse-associated symptoms and their treatment]. Urologie. 2024 Jan;63(1):43-50. doi: 10.1007/s00120-023-02247-6. Epub 2023 Dec 28. German. PMID 38153429
- [Derived] Himmler M, Gottl K, Witczak M, Yassouridis A, Gold DM, Liedl B. The impact of transvaginal, mesh-augmented level one apical repair on anorectal dysfunction due to pelvic organ prolapse. Int Urogynecol J. 2022 Nov;33(11):3261-3273. doi: 10.1007/s00192-022-05151-3. Epub 2022 Mar 28. PMID 35347368
- See also: AMS website — http://www.americanmedicalsystems.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phases duration:
  Phase I: May 2006 - Oct 2009 Phase II: Feb 2007 - Jun 2010 Phase III/IV: Apr 2007 - May 2010 Phase V: Apr 2008 - Jan 2011 Phase VI: Oct 2008 - Mar 2010 Phase VII: Apr 2009 - Feb 2012
Pre-assignment Details: Only those subjects who meet all study criteria, provide written consent and are implanted with an AMS PFR System device for prolapse repair will be considered evaluable for analysis in the study
Groups:
- Phase I (IntePro, US Only): AMS Apogee™ with IntePro: Mesh for the treatment of posterior vaginal wall prolapse
- Phase I (Intexen LP, US Only): AMS Apogee™ with InteXen LP: Graft for the treatment of posterior vaginal wall prolapse
- Phase II (France Only): AMS Perigee™ with IntePro: Mesh for the treatment of anterior vaginal wall prolapse.
- Phase III/IV (Perigee IntePro Lite, US Only): AMS Perigee™ with IntePro Lite: Mesh for the treatment of anterior vaginal wall prolapse Subjects in Phases III and IV were to be implanted with either an Apogee with IntePro Lite device, a Perigee with IntePro Lite device, or both devices
- Phase III/IV (Apogee IntePro Lite, US Only): AMS Apogee™ with IntePro Lite: Mesh for the treatment of posterior vaginal wall prolapse Subjects in Phases III and IV were to be implanted with either an Apogee with IntePro Lite device, a Perigee with IntePro Lite device, or both devices
- Phase V (Elevate Posterior IntePro Lite, US & EU): AMS Elevate™ Apical & Posterior with IntePro Lite: Mesh for the treatment of apical & posterior vaginal wall prolapse
- Phase V (Elevate Posterior InteXen LP, US Only): AMS Elevate™ Apical & Posterior with InteXen LP: Graft for the treatment of apical & posterior vaginal wall prolapse
- Phase VI (Elevate Anterior Gen 1, for Study Use Only, EU Only): AMS Elevate™ Anterior & Apical with IntePro Lite: Mesh for the treatment of anterior & apical vaginal wall prolapse (Generation 1, for PROPEL study use only)
- Phase VII (Elevate Anterior Gen 2, US & EU): AMS Elevate™ Anterior & Apical with IntePro Lite: Mesh for the treatment of anterior & apical vaginal wall prolapse (Generation 2)
Period: Overall Study
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, for Study Use Only, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Started | 141 | 26 | 81 | 56 | 55 | 139 | 23 | 35 | 142
Completed | 110 | 23 | 63 (Ph-II ended before all subjects had 24M b/c Perigee next generation was already under trial P-III/IV) | 46 | 42 | 113 | 23 | 34 (Ph-VI ended after 12M b/c next generation of Elevate Anterior was already under trial in Phase VII) | 124
Not Completed | 31 | 3 | 18 | 10 | 13 | 26 | 0 | 1 | 18
Not completed — Lost to Follow-up | 31 | 3 | 18 | 10 | 13 | 26 | 0 | 1 | 18

BASELINE CHARACTERISTICS:
Groups:
- Phase VI (Elevate Anterior Gen 1, EU Only): AMS Elevate™ Anterior & Apical with IntePro Lite: Mesh for the treatment of anterior & apical vaginal wall prolapse (Generation 1, For PROPEL Study Use Only)
- Total: Total of all reporting groups
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU) | Total
Number analyzed (Participants) | 141 | 26 | 81 | 56 | 55 | 139 | 23 | 35 | 142 | 698
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (12.2) | 63.4 (9.0) | 69.7 (10.9) | 63.4 (11.1) | 63.3 (11.8) | 62.5 (11.6) | 63.4 (9.6) | 65.4 (8.4) | 63.9 (9.8) | NA (0) — Mean age of the cohort was not analyzed and access to the database to calculate mean age for total is no longer available.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 26 | 81 | 56 | 55 | 139 | 23 | 35 | 142 | 698
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With an ICS (International Incontinence Society) POP-Q (Pelvic Organ Prolapse Quantification System) Stage of </= Stage I in the Posterior Compartment at One Year Post Procedure
Description: Analysis includes only subjects with posterior vaginal wall prolapse >= stage II at baseline. The POP-Q primary endpoint analysis employed the last observed failure carried forward method. Subjects with a follow-up POP-Q stage ≥ stage II were counted as failures, whereas subjects with a follow-up POP-Q stage < stage I were counted as successes. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a failure were counted as failures. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a success were counted as missing. Exact 95% confidence intervals were calculated via binomial distribution and were limited to subjects having a POPQ ≥ stage II at baseline.
Time Frame: 12-months
Population: Analysis conducted only for those subjects with posterior vaginal wall prolapse >= stage II at baseline. Where a "zero" is indicated, no subjects meeting this criteria were enrolled.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 117 | 24 | 0 | 0 | 44 | 120 | 23 | 0 | 0
percentage of participant | 93.2 [87.0 to 97.0] | 100 [85.8 to 100] |  |  | 93.2 [81.3 to 98.6] | 92.5 [86.2 to 96.5] | 100 [85.2 to 100] |  |

2. Secondary Outcome: QoL Status - Defined as the Improvement in Subjects' QoL Over Baseline Values as Measured in Three Questionnaires Post Procedure: PISQ-12
Description: Quality of Life as measure by Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). A higher or increasing score represents an improvement in perceived sexual function versus baseline.
  Changes in QoL scores between follow-up and baseline were presented. Only those subjects who completed both baseline and follow-up were included.
Time Frame: 6 Months
Population: Changes in QoL scores between follow-up and baseline were presented. Only those subjects who completed both baseline and follow-up were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 67 | 8 | 24 | 16 | 18 | 47 | 9 | 16 | 51
scores on a scale
  PISQ-12 mean score at baseline | 32.5 (7.1) | 32.1 (5.6) | 34.8 (5.5) | 33.4 (5.6) | 32.4 (6.4) | 34.0 (5.9) | 33.9 (4.4) | 34.0 (4.8) | 32.6 (8.1)
  PISQ-12 mean score at 6M | 37.1 (5.7) | 36.8 (7.2) | 36.8 (4.7) | 35.4 (5.9) | 35.4 (5.9) | 36.3 (5.5) | 35.0 (7.7) | 38.1 (6.4) | 36.6 (6.1)

3. Secondary Outcome: Procedural Time
Description: Procedural time was measured as the time between the first incision to place the study device and the time to close the vaginal incision for the study device. Procedure duration in minutes
Time Frame: Approximately 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 141 | 26 | 81 | 56 | 55 | 139 | 23 | 35 | 142
minutes | 44.8 (20.3) | 40.8 (17.7) | 50.2 (38.3) | 42.4 (16.4) | 51.7 (23.1) | 45.8 (19.2) | 48.6 (14.8) | 63.5 (19.0) | 54.6 (21.5)

4. Secondary Outcome: Estimated Blood Loss
Description: Estimated Blood Loss - defined as the estimated blood loss associated with the implantation of the study device, measured in ml
Time Frame: Approximately 30 minutes
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 139 | 26 | 80 | 56 | 55 | 139 | 23 | 35 | 142
milliliters | 68.6 (67.8) | 67.7 (43.9) | 48.8 (29.3) | 58.4 (54.7) | 58.9 (44.6) | 55.4 (45.7) | 62.4 (39.0) | 84.4 (60.9) | 75.5 (76.3)

5. Secondary Outcome: Percent of Subjects Experiencing Major Device Related Complications
Description: This may have included: perforation of internal organs during the implant procedure; graft erosion; serious infection requiring intravenous antibiotics; death, related to procedure or device; blood loss related to device placement which may have required blood transfusion during the procedure
Time Frame: Through 24 months
Population: Total subjects experienced major complications(%)
Measure: Number; unit: Percentage of participants
Groups:
- Phase II (France Only): AMS Perigee™ with IntePro: Mesh for the treatment of anterior vaginal wall prolapse.
  Phase II ended before all subjects reached their 24M follow up visit because next generation of Perigee was already under trial in Phase III/IV
- Phase VI (Elevate Anterior Gen 1, EU Only): AMS Elevate™ Anterior & Apical with IntePro Lite: Mesh for the treatment of anterior & apical vaginal wall prolapse (Generation 1, For PROPEL Study Use Only) Phase VI ended after 12M visit because next generation of Elevate Anterior was already under trial in Phase VII
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 141 | 26 | 81 | 56 | 55 | 139 | 23 | 35 | 142
Percentage of participants
  Perforation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Graft erosion | 0.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious infe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Death related to procedure or device | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood loss | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.7

6. Secondary Outcome: Rate of Graft Extrusions
Description: Rate of Graft Extrusion pertains to study device graft exposure/protrusion through the vaginal wall
Time Frame: Through 24 months
Population: Rate of subjects experiencing graft exposure through the vagina (%)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 141 | 26 | 81 | 56 | 55 | 139 | 23 | 35 | 142
Percentage of participants | 9.2 | 0 | 3.7 | 5.4 | 7.3 | 7.9 | 0 | 5.7 | 5.6

7. Secondary Outcome: Rates of de Novo or Worsening Urinary and/or Anal Incontinence
Description: Rate of subjects experiencing de novo or worsening urinary and or/ anal incontinence
Time Frame: Through 24 months
Population: Rate of subjects experiencing different type of incontinenece (%)
Measure: Number; unit: Percentage of participants
Groups:
- Phase II (France Only): AMS Perigee™ with IntePro: Mesh for the treatment of anterior vaginal wall prolapse.
  Phase II ended before all subjects had their 24M visit because next generation of Perigee was already under trial in Phase III/IV
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 141 | 26 | 81 | 56 | 55 | 139 | 23 | 35 | 142
Percentage of participants
  Urinary Incontinence - de novo Stress | 0 | 3.8 | 12.3 | 1.8 | 0 | 0 | 0 | 11.4 | 4.2
  Urinary Incontinence - worsening Stress | 0 | 0 | 8.6 | 0 | 0 | 0.7 | 0 | 11.4 | 0
  Urinary Incontinence - de novo Urge | 0 | 0 | 1.2 | 1.8 | 1.8 | 0 | 0 | 0 | 0.7
  Urinary Incontinence - Worsening Urge | 0 | 0 | 0 | 1.8 | 0 | 0 | 4.3 | 2.9 | 0.7
  Urinary Incontinence - de novo Mixed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2.9 | 0
  Urinary Incontinence - Worsening Mixed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2.9 | 0.7
  Fecal Incontinence | 0 | 0 | 0 | 0 | 0 | 0.7 | 0 | 0 | 0

8. Secondary Outcome: Wong-Baker Faces Pain Scale at 6 Weeks Post Procedure
Description: Pain - defined as the level of pain or discomfort associated with the pelvic area measured by the Wong-Baker Faces Pain Scale (scale of 0-10, with 10 indicating "hurts worst") at baseline, and 6 weeks post procedure
Time Frame: baseline and 6 weeks
Population: Changes in pain scores between follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 136 | 25 | 79 | 55 | 53 | 134 | 22 | 34 | 140
scores on a scale
  Mean level of pain per WBPS at baseline | 1.9 (2.5) | 2.0 (2.2) | 1.5 (1.8) | 1.2 (2.1) | 1.4 (2.1) | 1.8 (2.2) | 2.1 (2.9) | 1.1 (1.5) | 1.4 (2.0)
  Mean level of pain per WBPS at 6 weeks post-op | 0.7 (1.3) | 0.2 (0.6) | 0.9 (1.5) | 0.5 (1.1) | 0.7 (1.4) | 0.6 (1.3) | 0.8 (1.4) | 0.5 (1.0) | 0.7 (1.3)

9. Secondary Outcome: Patient Satisfaction Questionnaire at 6 Months by Question (Q#1)
Description: Subject satisfaction with experience and outcomes of the procedure, as reported on the Patient Satisfaction Questionnaires at 6 months post-procedure.
Time Frame: 6 Months
Population: Overall, what outcome do you feel you have achieved after having this surgery? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Groups:
- Phase V (Elevate Posterior InteXen LP, US & Only): AMS Elevate™ Apical & Posterior with InteXen LP: Graft for the treatment of apical & posterior vaginal wall prolapse
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US & Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 129 | 26 | 73 | 47 | 46 | 131 | 23 | 34 | 131
Percentage of participants
  Did not answer this question | 0.8 | 0 | 5.5 | 0 | 0 | 2.3 | 0 | 2.9 | 0.8
  Worse than before surgery | 0 | 0 | 0 | 4.3 | 2.2 | 1.5 | 0 | 2.9 | 1.5
  No improvement from before surgery | 0 | 0 | 0 | 0 | 0 | 0.8 | 0 | 0 | 1.5
  Some improvement from before surgery | 17.1 | 15.4 | 8.2 | 21.3 | 8.7 | 21.4 | 13.0 | 11.8 | 12.2
  A lot of improvement from before surgery | 82.2 | 84.6 | 86.3 | 74.5 | 89.1 | 74.0 | 87.0 | 82.4 | 84.0

10. Secondary Outcome: Surgical Revision Rate
Description: The monitoring of AEs occured through the end of the follow up period. Any continuing AEs past the 24M visit or early exit of subject was not followed to resolution.
Time Frame: Through 24 months
Population: Percentage of total subjects experienced surgical revision (%)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 141 | 26 | 81 | 56 | 55 | 139 | 23 | 35 | 142
Percentage of participants | 7.1 | 0 | 11.1 | 5.4 | 3.6 | 8.6 | 4.3 | 25.7 | 9.2

11. Secondary Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I at 6 Months
Description: The POP-Q primary endpoint analysis employed the last observed failure carried forward method. Subjects with a follow-up POP-Q stage ≥ stage II were counted as failures, whereas subjects with a follow-up POP-Q stage < stage I were counted as successes. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a failure were counted as failures. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a success were counted as missing. Exact 95% confidence intervals were calculated via binomial distribution and were limited to subjects having a POPQ ≥ stage II at baseline.
Time Frame: 6 months
Population: POP-Q analysis employed last failure carried forward method, which carries subject's objective failure at previous visits if the results are missing in the visit of interest. It's also considers re-operation for recurrent in study compartment as failure. 95% CI calculated via binominal distribution including only subjects w/POP-Q≥II at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 125 | 26 | 73 | 47 | 46 | 126 | 23 | 34 | 131
Percentage of participants
  Posterior Compartment Success | 94.4 [88.8 to 97.7] | 100 [86.8 to 100] | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | 91.3 [79.2 to 97.6] | 96.8 [92.1 to 99.1] | 100 [85.2 to 100] | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment
  Apical Compartment Success | 94.7 [82.3 to 99.4] | 100 [59.0 to 100] | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | 100 [66.4 to 100] | 92.5 [79.6 to 98.4] | 90.9 [58.7 to 99.8] | 90.0 [73.5 to 97.9] | 98.8 [93.4 to 100]
  Anterior Compartment Success | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | 76.7 [65.4 to 85.8] | 91.5 [79.6 to 97.6] | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | 61.8 [43.6 to 77.8] | 86.3 [79.2 to 91.6]

12. Secondary Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I at 24 Months
Description: The POP-Q primary endpoint analysis employed the last observed failure carried forward method. Subjects with a follow-up POP-Q stage ≥ stage II were counted as failures, whereas subjects with a follow-up POP-Q stage < stage I were counted as successes. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a failure were counted as failures. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a success were counted as missing. Exact 95% confidence intervals were calculated via binomial distribution and were limited to subjects having a POPQ ≥ stage II at baseline.
  Note:
  1. Phase VI ended after 12M follow up visit because the next generation of the study device was already under clinical evaluation in Phase VII
  2. Phase II ended early before all subjects reached their 24M visit because the study device is no longer marketed due to release of models with enhancements to the design
Time Frame: 24 months
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 108 | 23 | 68 | 46 | 44 | 106 | 23 | 0 | 125
Percentage of participants
  Posterior Compartment Success | 93.5 [87.1 to 97.4] | 95.7 [78.1 to 99.9] | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | 90.9 [78.3 to 97.5] | 91.5 [84.5 to 96.0] | 90.9 [58.7 to 99.8] |  | NA [NA to NA] — Phase device does not treat this compartment
  Apical Compartment Success | 84.4 [67.2 to 94.7] | 100 [54.1 to 100] | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | 75.0 [42.1 to 99.6] | 88.2 [72.5 to 96.7] | 100 [85.2 to 100] |  | 96.2 [89.3 to 99.2]
  Anterior Compartment Success | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | 69.1 [56.7 to 79.8] | 87.0 [73.7 to 95.1] | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment | NA [NA to NA] — Phase device does not treat this compartment |  | 81.6 [73.7 to 88.0]

13. Secondary Outcome: Patient Satisfaction Questionnaire at 12 Months by Question (Q#1)
Description: as for outcome 9
Time Frame: 12 months
Population: Overall, what outcome do you feel you have achieved after having this surgery? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 119 | 24 | 71 | 45 | 44 | 126 | 23 | 34 | 125
Percentage of participants
  Did not answer this question | 0 | 4.2 | 7.0 | 0 | 0 | 1.6 | 0 | 2.9 | 0
  Worse than before surgery | 1.7 | 0 | 0 | 0 | 0 | 1.6 | 0 | 0 | 0.8
  No improvement from before surgery | 0 | 4.2 | 0 | 0 | 2.3 | 2.4 | 0 | 0 | 2.4
  Some improvement from before surgery | 17.6 | 12.5 | 14.1 | 13.3 | 4.5 | 23.0 | 26.1 | 8.8 | 6.4
  A lot of improvement from before surgery | 80.7 | 79.2 | 78.9 | 86.7 | 93.2 | 71.4 | 73.9 | 88.2 | 90.4

14. Secondary Outcome: Patient Satisfaction Questionnaire at 24 Months by Question (Q#1)
Description: Subject satisfaction with experience and outcomes of the procedure, as reported on the Patient Satisfaction Questionnaires at 6 months post-procedure.
  Note:
  1. Phase VI ended after 12M follow up visit because the next generation of the study device was already under clinical evaluation in Phase VII
  2. Phase II ended early before all subjects reached their 24M visit because the study device is no longer marketed due to release of models with enhancements to the design
Time Frame: 24 months
Population: Overall, what outcome do you feel you have achieved after having this surgery? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 110 | 23 | 63 | 46 | 42 | 113 | 23 | 0 | 124
Percentage of participants
  Did not answer this question | 0 | 4.3 | 11.1 | 2.2 | 0 | 0.9 | 0 |  | 0.8
  Worse than before surgery | 2.7 | 0 | 0 | 4.3 | 2.4 | 4.4 | 0 |  | 0.8
  No improvement from before surgery | 0.9 | 0 | 0 | 0 | 0 | 3.5 | 0 |  | 1.6
  Some improvement from before surgery | 10.9 | 4.3 | 7.9 | 17.4 | 11.9 | 20.4 | 30.4 |  | 12.1
  A lot of improvement from before surgery | 85.5 | 91.3 | 81.0 | 76.1 | 85.7 | 70.8 | 69.6 |  | 84.7

15. Secondary Outcome: Patient Satisfaction Questionnaire at 6 Months by Question (Q#2)
Description: as for outcome 9
Time Frame: 6 months
Population: How satisfied are you with the outcome of your prolapse surgery? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 129 | 26 | 73 | 47 | 46 | 131 | 23 | 34 | 131
Percentage of participants
  Did not answer this question | 0.8 | 0 | 5.5 | 0 | 0 | 2.3 | 0 | 0 | 0.8
  Not at all satisfied | 0.8 | 0 | 0 | 0 | 0 | 1.5 | 0 | 2.9 | 3.1
  Slightly satisfied | 0.8 | 3.8 | 0 | 2.1 | 2.2 | 4.6 | 0 | 2.9 | 1.5
  Moderately satisfied | 11.6 | 3.8 | 6.8 | 6.4 | 4.3 | 12.2 | 0 | 5.9 | 5.3
  Very satisfied | 34.1 | 38.5 | 47.9 | 46.8 | 34.8 | 38.2 | 47.8 | 61.8 | 40.5
  Extremely satisfied | 51.9 | 53.8 | 39.7 | 44.7 | 58.7 | 41.2 | 52.2 | 26.5 | 48.9

16. Secondary Outcome: Patient Satisfaction Questionnaire at 12 Months by Question (Q#2)
Description: Subject satisfaction with experience and outcomes of the procedure, as reported on the Patient Satisfaction Questionnaires at 12 months post-procedure.
Time Frame: 12 months
Population: How satisfied are you with the outcome of your prolapse surgery? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 119 | 24 | 71 | 45 | 44 | 126 | 23 | 34 | 125
Percentage of participants
  Did not answer this question | 0 | 4.2 | 7.0 | 0 | 0 | 0.8 | 0 | 2.9 | 0
  Not at all satisfied | 0.8 | 0 | 0 | 0 | 0 | 2.4 | 0 | 0 | 0.8
  Slightly satisfied | 4.2 | 4.2 | 0 | 0 | 2.3 | 2.4 | 8.7 | 0 | 4.8
  Moderately satisfied | 13.4 | 8.3 | 9.9 | 17.8 | 6.8 | 13.5 | 4.3 | 8.8 | 3.2
  Very satisfied | 32.8 | 33.3 | 45.1 | 40 | 40.9 | 42.1 | 26.1 | 52.9 | 32.8
  Extremely satisfied | 48.7 | 50 | 38.0 | 42.2 | 50.0 | 38.9 | 60.9 | 35.3 | 58.4

17. Secondary Outcome: Patient Satisfaction Questionnaire at 24 Months by Question (Q#2)
Description: Subject satisfaction with experience and outcomes of the procedure, as reported on the Patient Satisfaction Questionnaires at 24 months post-procedure.
  Note:
  1. Phase VI ended after 12M follow up visit because the next generation of the study device was already under clinical evaluation in Phase VII
  2. Phase II ended early before all subjects reached their 24M visit because the study device is no longer marketed due to release of models with enhancements to the design
Time Frame: 24 months
Population: How satisfied are you with the outcome of your prolapse surgery? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 110 | 23 | 63 | 46 | 42 | 113 | 23 | 0 | 124
Percentage of participants
  Did not answer this question | 0 | 4.3 | 11.1 | 2.2 | 0 | 0.9 | 0 |  | 0.8
  Not at all satisfied | 3.6 | 0 | 0 | 4.3 | 2.4 | 2.7 | 0 |  | 2.4
  Slightly satisfied | 1.8 | 0 | 0 | 2.2 | 4.8 | 8.0 | 0 |  | 3.2
  Moderately satisfied | 11.8 | 4.3 | 6.3 | 8.7 | 9.5 | 9.7 | 8.7 |  | 5.6
  Very satisfied | 23.6 | 26.1 | 44.4 | 41.3 | 35.7 | 40.7 | 47.8 |  | 29.8
  Extremely satisfied | 59.1 | 65.2 | 38.1 | 41.3 | 47.6 | 38.1 | 43.5 |  | 58.1

18. Secondary Outcome: Patient Satisfaction Questionnaire at 6 Months by Question (Q#3)
Description: as for outcome 9
Time Frame: 6 months
Population: Would you recommend this procedure to a friend suffering from prolapse? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 129 | 26 | 73 | 47 | 46 | 131 | 23 | 34 | 131
Percentage of participants
  Did not answer this question | 2.3 | 0 | 5.5 | 0 | 0 | 2.3 | 0 | 0 | 0.8
  Yes | 94.6 | 100 | 94.5 | 95.7 | 93.5 | 96.9 | 100 | 97.1 | 96.9
  No | 3.1 | 0 | 0 | 4.3 | 6.5 | 0.8 | 0 | 2.9 | 2.3

19. Secondary Outcome: Patient Satisfaction Questionnaire at 12 Months by Question (Q#3)
Description: as for outcome 16
Time Frame: 12 months
Population: Would you recommend this procedure to a friend suffering from prolapse? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 119 | 24 | 71 | 45 | 44 | 126 | 23 | 34 | 125
Percentage of participants
  Did not answer this question | 1.7 | 4.2 | 7.0 | 0 | 0 | 2.4 | 0 | 5.9 | 1.6
  Yes | 92.4 | 95.8 | 93.0 | 100 | 97.7 | 96.0 | 95.7 | 94.1 | 96.8
  No | 5.9 | 0 | 0 | 0 | 2.3 | 1.6 | 4.3 | 0 | 1.6

20. Secondary Outcome: Patient Satisfaction Questionnaire at 24 Months by Question (Q#3)
Description: as for outcome 17
Time Frame: 24 months
Population: Would you recommend this procedure to a friend suffering from prolapse? (% of subjects answering this question)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 110 | 23 | 63 | 46 | 42 | 113 | 23 | 0 | 124
Percentage of participants
  Did not answer this question | 0.9 | 4.3 | 11.1 | 2.2 | 0 | 0.9 | 0 |  | 2.4
  Yes | 90.9 | 95.7 | 87.3 | 93.5 | 95.2 | 92.0 | 95.7 |  | 94.4
  No | 8.2 | 0 | 1.6 | 4.3 | 4.8 | 7.1 | 4.3 |  | 3.2

21. Secondary Outcome: Wong-Baker Faces Pain Scale at 3 Months Post Procedure
Description: Pain - defined as the level of pain or discomfort associated with the pelvic area measured by the Wong-Baker Faces Pain Scale at baseline and 3 months post procedure
Time Frame: baseline and 3 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 134 | 25 | 77 | 37 | 38 | 123 | 23 | 33 | 131
Percentage of participants
  Mean level of pain per WBPS at baseline | 1.9 (2.5) | 2.0 (2.2) | 1.5 (1.8) | 1.2 (2.2) | 1.6 (2.2) | 1.7 (2.0) | 2.2 (2.8) | 1.2 (1.5) | 1.4 (2.0)
  Mean level of pain per WBPS at 3 months post-op | 0.5 (1.0) | 0.2 (0.6) | 0.9 (1.5) | 0.2 (0.6) | 0.2 (0.6) | 0.3 (0.9) | 0.4 (0.8) | 0.4 (1.0) | 0.5 (1.2)

22. Secondary Outcome: QoL Status - Defined as the Improvement in Subjects' QoL Over Baseline Values as Measured in Three Questionnaires Post Procedure: PISQ-12
Description: Quality of Life as measure by Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). QoL scores for follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented.
Time Frame: 12 months
Population: QoL scores for follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented.
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 62 | 9 | 22 | 15 | 15 | 48 | 9 | 18 | 48
Percentage of participants
  PISQ-12 mean score at baseline | 33.4 (7.3) | 31.7 (5.4) | 35.3 (5.3) | 32.8 (5.5) | 33.0 (6.2) | 34.1 (6.1) | 34.3 (4.5) | 33.4 (4.8) | 31.9 (8.4)
  PISQ-12 mean score at 12M | 37.2 (5.9) | 33.8 (9.3) | 36.3 (4.9) | 34.9 (5.6) | 36.4 (5.8) | 36.5 (5.5) | 35.6 (5.5) | 37.7 (5.8) | 37.4 (5.7)

23. Secondary Outcome: QoL Status - Defined as the Improvement in Subjects' QoL Over Baseline Values as Measured in Three Questionnaires Post Procedure: PISQ-12
Description: Quality of Life as measure by Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) QoL scores for follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented.
Time Frame: baseline and 24 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 56 | 9 | 22 | 16 | 13 | 37 | 8 | 0 | 45
Percentage of participants
  PISQ-12 mean score at baseline | 32.4 (7.4) | 31.7 (5.4) | 34.5 (6.5) | 32.4 (5.3) | 31.9 (5.2) | 34.9 (5.8) | 33.6 (4.2) |  | 32.0 (8.4)
  PISQ-12 mean score at 24M | 36.9 (6.4) | 36.6 (5.3) | 36.0 (4.4) | 35.3 (4.6) | 35.9 (4.8) | 36.6 (6.5) | 34.6 (5.5) |  | 36.3 (6.1)

24. Secondary Outcome: QoL Status - Defined as the Improvement in Subjects' QoL Over Baseline Values as Measured in Three Questionnaires Post Procedure: PFIQ-7 at 6M
Description: Quality of Life as measure by Pelvic Floor Impact Questionnaire - Short Form 7(PFIQ-7) QoL scores for follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented. .
Time Frame: baseline and 6 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 124 | 25 | 65 | 47 | 45 | 123 | 23 | 30 | 127
Percentage of participants
  PFIQ-7 mean score at baseline | 70.4 (72.2) | 68.2 (62.8) | 54.9 (55.7) | 61.5 (75.7) | 58.9 (70.1) | 65.4 (59.8) | 60.2 (40.0) | 71.4 (67.2) | 59.8 (61.1)
  PFIQ-7 mean score at 6M | 16.3 (35.7) | 21.7 (44.0) | 9.9 (21.1) | 8.4 (20.5) | 9.2 (28.3) | 22.3 (40.8) | 6.0 (13.6) | 22.8 (36.5) | 12.9 (29.0)

25. Secondary Outcome: QoL Status - Defined as the Improvement in Subjects' QoL Over Baseline Values as Measured in Three Questionnaires Post Procedure: PFIQ-7 at 12M
Description: Quality of Life as measure by Pelvic Floor Impact Questionnaire - Short Form 7(PFIQ-7) QoL scores for follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented.
Time Frame: baseline and 12 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 117 | 22 | 67 | 45 | 42 | 120 | 23 | 28 | 122
Percentage of participants
  PFIQ-7 mean score at baseline | 64.9 (70.5) | 59.3 (48.2) | 59.1 (57.4) | 61.7 (74.6) | 57.5 (65.0) | 65.6 (59.7) | 60.2 (40.0) | 73.0 (68.1) | 55.8 (60.5)
  PFIQ-7 mean score at 12M | 13.1 (27.8) | 10.0 (19.8) | 9.1 (16.0) | 10.7 (21.8) | 8.8 (26.7) | 17.9 (39.9) | 8.5 (17.3) | 8.7 (13.6) | 14.0 (39.0)

26. Secondary Outcome: QoL Status - Defined as the Improvement in Subjects' QoL Over Baseline Values as Measured in Three Questionnaires Post Procedure: PFIQ-7 at 24M
Description: as for outcome 25
Time Frame: baseline and 24 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 108 | 21 | 55 | 45 | 41 | 108 | 23 | 0 | 121
Percentage of participants
  PFIQ-7 mean score at baseline | 59.1 (63.8) | 55.6 (46.0) | 60.9 (59.3) | 56.5 (71.6) | 59.0 (69.5) | 64.3 (56.5) | 60.2 (40.0) |  | 54.8 (56.1)
  PFIQ-7 mean score at 24M | 15.8 (40.9) | 5.0 (8.0) | 11.9 (27.8) | 10.5 (36.1) | 7.8 (23.4) | 17.9 (34.7) | 9.7 (15.0) |  | 9.3 (24.8)

27. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI (Pelvic Floor Distress Inventory) Sub-scale UDI (Urinary Distress Inventory) at 6M
Description: Quality of Life as measure by PFDI subscale UDI. UDI scale ranges from 0-100 with 100 representing the most urinary distress. Changes in UDI scores between follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented.
Time Frame: baseline and 6 months
Population: Changes in QoL scores between follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 128 | 26 | 64 | 46 | 45 | 130 | 23 | 34 | 130
scores on a scale
  PFDI- UDI mean score at baseline | 98.4 (59.6) | 106.7 (63.4) | 65.5 (34.5) | 93.2 (55.1) | 93.0 (55.0) | 97.6 (59.8) | 83.0 (40.4) | 75.5 (54.2) | 87.0 (55.5)
  PFDI- UDI mean score at 6M | 29.1 (37.2) | 36.4 (38.4) | 15.4 (19.1) | 21.8 (22.4) | 29.2 (37.7) | 31.2 (35.6) | 14.6 (23.4) | 29.7 (33.5) | 23.2 (27.2)

28. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI Sub-scale UDI (Urinary Distress Inventory) at 12M
Description: Quality of Life as measure by Pelvic Floor Distress Inventory(PFDI). PFDI assesses the impact of urinary, prolapse and colorectal distress at baseline and post-op. QoL scores for follow-up and baseline were presented. Only data from those subjects who completed both baseline and follow-up were presented.
Time Frame: baseline and 12 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 119 | 24 | 63 | 45 | 44 | 126 | 23 | 34 | 125
Percentage of participants
  PFDI- UDI mean score at baseline | 97.5 (59.1) | 103.6 (53.1) | 66.7 (33.7) | 92.4 (51.7) | 93.4 (54.4) | 97.6 (58.6) | 83.0 (40.4) | 75.5 (54.2) | 84.4 (50.8)
  PFDI- UDI mean score at 12M | 34.8 (44.3) | 28.3 (40.7) | 14.0 (14.6) | 22.8 (25.4) | 20.3 (28.9) | 33.0 (36.5) | 19.8 (22.6) | 26.4 (30.8) | 21.0 (28.1)

29. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI Sub-scale UDI (Urinary Distress Inventory) at 24M
Description: as for outcome 28
Time Frame: baseline and 24 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 110 | 22 | 55 | 45 | 42 | 113 | 23 | 0 | 124
Percentage of participants
  PFDI- UDI mean score at baseline | 96.5 (56.7) | 94.9 (55.8) | 69.9 (34.5) | 89.6 (51.5) | 95.8 (56.9) | 97.6 (57.1) | 83.0 (40.4) |  | 82.5 (50.6)
  PFDI- UDI mean score at 24M | 28.1 (35.7) | 13.2 (17.1) | 19.8 (22.7) | 20.3 (21.8) | 29.8 (39.1) | 29.4 (30.9) | 15.1 (14.1) |  | 20.5 (25.0)

30. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI Sub-scale POPDI (Pelvic Organ Prolapse Distress Inventory) at 6M
Description: as for outcome 28
Time Frame: baseline and 6 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 127 | 26 | 63 | 47 | 46 | 130 | 23 | 34 | 130
Percentage of participants
  PFDI- POPDI mean score at baseline | 137.0 (69.9) | 128.9 (65.9) | 102.3 (45.4) | 112.0 (67.2) | 115.7 (69.9) | 122.7 (64.3) | 115.5 (53.5) | 105.4 (61.3) | 107.8 (65.9)
  PFDI- POPDI mean score at 6M | 37.5 (43.4) | 34.7 (48.8) | 27.8 (34.8) | 19.1 (21.9) | 30.3 (35.2) | 42.9 (50.9) | 21.6 (24.4) | 36.1 (48.3) | 31.8 (40.7)

31. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI Sub-scale CRADI (Colo-Rectal-Anal Distress Inventory) at 6M
Description: as for outcome 28
Time Frame: baseline and 6 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 127 | 26 | 63 | 46 | 45 | 128 | 23 | 33 | 128
Percentage of participants
  PFDI- CRADI mean score at baseline | 129.6 (88.1) | 125.8 (83.3) | 52.6 (48.3) | 82.4 (75.1) | 94.1 (71.8) | 110.0 (74.0) | 102.1 (65.9) | 70.5 (60.7) | 80.6 (68.1)
  PFDI- CRADI mean score at 6M | 49.2 (63.1) | 45.3 (42.6) | 30.6 (38.9) | 23.4 (28.3) | 31.2 (36.5) | 52.9 (62.5) | 29.0 (35.6) | 41.8 (44.1) | 36.3 (46.5)

32. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI Sub-scale POPDI (Pelvic Organ Prolapse Distress Inventory) at 12M
Description: as for outcome 28
Time Frame: baseline and 12 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 119 | 24 | 62 | 45 | 44 | 126 | 23 | 34 | 124
Percentage of participants
  PFDI- POPDI mean score at baseline | 135.1 (68.9) | 128.2 (55.4) | 103.3 (45.6) | 105.7 (58.8) | 116.1 (65.9) | 122.0 (63.7) | 115.5 (53.5) | 105.4 (61.3) | 104.4 (62.6)
  PFDI- POPDI mean score at 12M | 45.2 (49.3) | 42.4 (50.5) | 25.8 (30.3) | 23.6 (30.3) | 19.9 (28.0) | 43.0 (52.5) | 29.9 (27.7) | 32.5 (34.2) | 23.8 (36.5)

33. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI Sub-scale POPDI (Pelvic Organ Prolapse Distress Inventory) at 24M
Description: as for outcome 28
Time Frame: baseline and 24 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Groups:
- Phase II (France Only): AMS Perigee™ with IntePro: Mesh for the treatment of anterior vaginal wall prolapse.
  Phase II ended before all subjects reached their 24M follow up visit because next generation of Perigee was already under trial in Phase III/IVmodels
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 109 | 22 | 54 | 45 | 42 | 113 | 23 | 0 | 124
Percentage of participants
  PFDI- POPDI mean score at baseline | 132.4 (68.3) | 113.2 (56.6) | 107.4 (46.3) | 104.7 (60.1) | 116.1 (65.1) | 121.7 (63.0) | 115.5 (53.5) |  | 103.3 (59.1)
  PFDI- POPDI mean score at 24M | 36.4 (48.9) | 13.8 (18.1) | 31.7 (37.6) | 23.8 (28.1) | 31.1 (36.7) | 37.6 (51.9) | 21.9 (21.6) |  | 24.8 (32.3)

34. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI Sub-scale CRADI (Colo-Rectal-Anal Distress Inventory) at 12M
Description: as for outcome 28
Time Frame: baseline and 12 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 119 | 24 | 63 | 44 | 43 | 126 | 23 | 33 | 121
Percentage of participants
  PFDI- CRADI mean score at baseline | 129.8 (88.9) | 123.5 (73.8) | 50.9 (49.3) | 85.1 (72.3) | 100.8 (72.8) | 108.2 (71.7) | 102.1 (65.9) | 70.5 (60.7) | 77.2 (66.9)
  PFDI- CRADI mean score at 12M | 46.6 (60.5) | 47.3 (51.2) | 27.3 (36.2) | 29.9 (42.1) | 22.7 (30.6) | 49.6 (55.1) | 32.5 (41.0) | 39.4 (42.8) | 29.4 (44.7)

35. Secondary Outcome: QoL Status - Improvement in Subjects' QoL Over Baseline Values as Measured by PFDI Sub-scale CRADI (Colo-Rectal-Anal Distress Inventory) at 24M
Description: as for outcome 28
Time Frame: baseline and 24 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 109 | 22 | 54 | 45 | 42 | 112 | 23 | 0 | 122
Percentage of participants
  PFDI- CRADI mean score at baseline | 126.9 (84.9) | 110.6 (73.2) | 58.3 (50.4) | 79.8 (73.2) | 95.5 (74.3) | 105.9 (70.3) | 102.1 (65.9) |  | 77.2 (65.2)
  PFDI- CRADI mean score at 24M | 40.2 (53.5) | 22.0 (30.6) | 33.7 (41.3) | 25.1 (38.5) | 27.2 (37.8) | 42.7 (52.7) | 29.4 (36.7) |  | 28.9 (35.3)

36. Primary Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I in the Apical Compartment at One Year Post Procedure
Description: Analysis includes only subjects with uterine descent >= stage II at baselineThe POP-Q primary endpoint analysis employed the last observed failure carried forward method. Subjects with a follow-up POP-Q stage ≥ stage II were counted as failures, whereas subjects with a follow-up POP-Q stage < stage I were counted as successes. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a failure were counted as failures. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a success were counted as missing. Exact 95% confidence intervals were calculated via binomial distribution and were limited to subjects having a POPQ ≥ stage II at baseline.
Time Frame: 12-months
Population: Analysis includes only subjects with uterine descent >=stage II at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 36 | 7 | 0 | 0 | 7 | 37 | 11 | 30 | 73
percentage of participant | 86.1 [70.5 to 95.3] | 100 [59.0 to 100] |  |  | 100 [59.0 to 100] | 89.2 [74.6 to 97.0] | 90.9 [58.7 to 100] | 90.0 [73.5 to 97.9] | 95.9 [88.5 to 99.1]

37. Primary Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I in the Anterior Compartment at One Year Post Procedure
Description: Analysis includes only subjects with anterior vaginal wall prolapse >= stage II at baseline. The POP-Q primary endpoint analysis employed the last observed failure carried forward method (LFCF). Subjects with a follow-up POP-Q stage ≥ stage II were counted as failures, whereas subjects with a follow-up POP-Q stage < stage I were counted as successes. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a failure were counted as failures. Subjects who missed the POP-Q at the visit of interest and had the previous visited noted as a success were counted as missing. Exact 95% confidence intervals were calculated via binomial distribution and were limited to subjects having a POPQ ≥ stage II at baseline.
Time Frame: 12-months
Population: Analysis includes only subjects with anterior vaginal wall prolapse >= stage II at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participant
Groups:
- Phase VI (Elevate Anterior Gen 1, EU Only): AMS Elevate™ Anterior & Apical with IntePro Lite: Mesh for the treatment of anterior & apical vaginal wall prolapse (Generation 1, Fot PROPEL Study Use Only)
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 0 | 0 | 73 | 44 | 0 | 0 | 0 | 34 | 127
percentage of participant |  |  | 71.2 [59.4 to 81.2] | 85.1 [71.7 to 93.8] |  |  |  | 58.8 [40.7 to 75.4] | 87.4 [80.3 to 92.6]

38. Secondary Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I in the Posterior Compartment at 6M Post Procedure
Description: as for outcome 1
Time Frame: 6 months
Population: Analysis includes only subjects with posterior vaginal wall prolapse >= stage II at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 125 | 26 | 0 | 0 | 46 | 126 | 23 | 0 | 0
percentage of participants | 94.4 [88.8 to 97.7] | 100 [86.8 to 100] |  |  | 91.3 [79.2 to 97.6] | 96.8 [92.1 to 99.1] | 100 [85.2 to 100] |  |

39. Secondary Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I in the Posterior Compartment at 24M Post Procedure
Description: as for outcome 1
Time Frame: 24 months
Population: Analysis includes only subjects with posterior vaginal wall prolapse >= stage II at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 108 | 23 | 0 | 0 | 44 | 106 | 23 | 0 | 0
percentage of participants | 93.5 [87.1 to 97.4] | 95.7 [78.1 to 99.9] |  |  | 90.9 [78.3 to 97.5] | 91.5 [84.5 to 96.0] | 100 [85.2 to 100] |  |

40. Other Pre Specified Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I in the Apical Compartment at 6M Post Procedure
Description: as for outcome 36
Time Frame: 6 months
Population: Analysis includes only subjects with uterine descent >=stage II at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 38 | 7 | 0 | 0 | 9 | 40 | 11 | 30 | 82
Percentage of participants | 94.7 [82.3 to 99.4] | 100 [59.0 to 100] |  |  | 100 [66.4 to 100] | 92.5 [79.6 to 98.4] | 90.9 [58.7 to 99.8] | 90.0 [73.5 to 97.9] | 98.8 [93.4 to 100]

41. Other Pre Specified Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I in the Apical Compartment at 24M Post Procedure
Description: as for outcome 36
Time Frame: 24 months
Population: Analysis includes only subjects with uterine descent >=stage II at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 32 | 6 | 0 | 0 | 7 | 34 | 11 | 0 | 79
Percentage of participants | 84.4 [67.2 to 94.7] | 100 [54.1 to 100] |  |  | 85.4 [42.1 to 99.6] | 88.2 [72.5 to 96.7] | 90.9 [58.7 to 99.8] |  | 96.2 [89.3 to 99.2]

42. Secondary Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I in the Anterior Compartment at 6M Post Procedure
Description: as for outcome 37
Time Frame: 6 months
Population: Analysis includes only subjects with anterior vaginal wall prolapse >= stage II at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 0 | 0 | 73 | 47 | 0 | 0 | 0 | 34 | 131
percentage of participants |  |  | 76.7 [65.4 to 85.8] | 91.5 [79.6 to 97.6] |  |  |  | 61.8 [43.6 to 77.8] | 86.3 [79.2 to 91.6]

43. Secondary Outcome: Percent of Subjects With an ICS POP-Q Stage of </= Stage I in the Anterior Compartment at 24M Post Procedure
Description: as for outcome 37
Time Frame: 24 months
Population: Analysis includes only subjects with anterior vaginal wall prolapse >= stage II at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Number analyzed (Participants) | 0 | 0 | 68 | 46 | 0 | 0 | 0 | 0 | 125
Percentage of participants |  |  | 69.1 [56.7 to 79.8] | 87.0 [73.7 to 95.1] |  |  |  |  | 81.6 [73.7 to 88.0]

ADVERSE EVENTS:
Time Frame: The monitoring of AEs occured through the end of the follow up period. Any continuing AEs past the 24M visit or early exit of subject was not followed to resolution.
Description: The Astora Women's Health business is closing and will no longer be able to provide updates to this results section. Specific adverse event data can no longer be provided or updated because the database that holds the raw data is no longer accessible by Astora personnel.
Arm/Group | Phase I (IntePro, US Only) | Phase I (Intexen LP, US Only) | Phase II (France Only) | Phase III/IV (Perigee IntePro Lite, US Only) | Phase III/IV (Apogee IntePro Lite, US Only) | Phase V (Elevate Posterior IntePro Lite, US & EU) | Phase V (Elevate Posterior InteXen LP, US Only) | Phase VI (Elevate Anterior Gen 1, EU Only) | Phase VII (Elevate Anterior Gen 2, US & EU)
Serious Adverse Events (participants affected / at risk) | 10/141 | 1/26 | 11/81 | 3/56 | 3/55 | 8/139 | 1/23 | 8/35 | 11/142
Other Adverse Events (participants affected / at risk) | 30/141 | 3/26 | 30/81 | 20/56 | 20/55 | 30/139 | 3/23 | 7/35 | 62/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (IntePro, US Only) (N=141) | Phase I (Intexen LP, US Only) (N=26) | Phase II (France Only) (N=81) | Phase III/IV (Perigee IntePro Lite, US Only) (N=56) | Phase III/IV (Apogee IntePro Lite, US Only) (N=55) | Phase V (Elevate Posterior IntePro Lite, US & EU) (N=139) | Phase V (Elevate Posterior InteXen LP, US Only) (N=23) | Phase VI (Elevate Anterior Gen 1, EU Only) (N=35) | Phase VII (Elevate Anterior Gen 2, US & EU) (N=142)
any Serious Adverse Event (General disorders) | 10 (10) | 1 (1) | 11 (11) | 3 (3) | 3 (3) | 8 (8) | 1 (1) | 8 (8) | 11 (11) — Serious Adverse Events are presented as a total. Breaking these SAEs out cannot be accomplished as the study database is not accessible. These SAEs are represented by multiple organ systems
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (IntePro, US Only) (N=141) | Phase I (Intexen LP, US Only) (N=26) | Phase II (France Only) (N=81) | Phase III/IV (Perigee IntePro Lite, US Only) (N=56) | Phase III/IV (Apogee IntePro Lite, US Only) (N=55) | Phase V (Elevate Posterior IntePro Lite, US & EU) (N=139) | Phase V (Elevate Posterior InteXen LP, US Only) (N=23) | Phase VI (Elevate Anterior Gen 1, EU Only) (N=35) | Phase VII (Elevate Anterior Gen 2, US & EU) (N=142)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 5 (5) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 8 (9) — Additional AEs not reported in the secondary endpoints
Dyspareunia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (7) — Additional AEs not reported in the secondary endpoints
Infection- Vaginal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) — Additional AEs not reported in the secondary endpoints
Device Malfunction (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Additional AEs not reported in the secondary endpoints
Any non-serious adverse events (General disorders) | 30 | 3 | 30 | 20 | 20 | 30 | 3 | 7 | 62 — why cant provide specific ae data? these numbers are a repeat of the data in the non-serious data table

LIMITATIONS AND CAVEATS:
1. Ph- II ended before all subjects reached 24M visit b/c the next generation of Perigee was already under trial, Ph-III/IV
2. Ph-VI ended after 12M visit because the next generation of study device was already under clinical evaluation in Phase VII

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less